CLINICAL TRIAL: NCT05844930
Title: Double Blinded Prospective Pilot Study to Determine the Safety and Effectiveness of a Connective Tissue Allograft (ActiveMatrix) vs. Standard of Care in Adhesive Capsulitis of the Shoulder
Brief Title: A Study to Determine the Safety and Effectiveness of a Connective Tissue Allograft (ActiveMatrix) Verses Standard of Care in Adhesive Capsulitis of the Shoulder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Skye Biologics, Inc. (Industry)
Responsible Party: Principal Investigator, Eric F Berkman, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-21-0706
Record Dates: First submitted 2023-04-21; First posted 2023-05-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Adhesive Capsulitis
Keywords: Frozen Shoulder; musculoskeletal injuries
MeSH Terms: conditions — Bursitis | interventions — Adrenal Cortex Hormones; Triamcinolone; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-articular Injection of Corticosteroid Plus Lidocaine (Active Comparator): Participants will receive a corticosteroid injection consisting of Triamcinolone 20 mg (1cc) with Lidocaine 10 mg/ml (5 cc).
  Interventions: Drug: Corticosteroid; Drug: Lidocaine
- Intra-articular Injection of ActiveMatrix Plus Lidocaine (Experimental): Participants will receive an injection consisting of ActiveMatrix (1cc; Skye Biologics, Inc.) with Lidocaine 10 mg/ml (5cc).
  Interventions: Other: ActiveMatrix; Drug: Lidocaine

INTERVENTIONS:
Drug: Corticosteroid — Triamcinolone 20 mg (1cc)
  Other Names: Triamcinolone
  Arms: Intra-articular Injection of Corticosteroid Plus Lidocaine
Other: ActiveMatrix — 1cc ActiveMatrix (Skye Biologics, Inc.)
  Other Names: Human Placental Connective Tissue-Derived Allograft
  Arms: Intra-articular Injection of ActiveMatrix Plus Lidocaine
Drug: Lidocaine — Lidocaine 10 mg/mL (5cc)

SUMMARY:
The purpose of this study is to compare ActiveMatrix® to standard of care corticosteroid injection in the treatment of adhesive capsulitis of the shoulder (frozen shoulder).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Have a clinical diagnosis of adhesive capsulitis, defined as: i. pain along the C5 dermatome; and ii. limitations of passive range of motion of more than 20 degrees in the abduction internal rotation, neutral external rotation, forward elevation and abduction planes when compared to the contralateral shoulder
* Have no contraindications or allergies to the treatment administered
* Have experienced shoulder pain for more than 6 weeks and less than 1 year (to ensure the patient is in the "freezing" stage of adhesive capsulitis).
* Have current imaging studies (plain radiographs and MRI exams) of the shoulder to rule out other etiologic diagnoses.

Exclusion Criteria:

* Any prior treatment for this episode of shoulder pain, such as prior intra-articular injection or prior physiotherapy
* Evidence, based on MRI or plain radiographs, of any pathology within the shoulder other than adhesive capsulitis (e.g., glenohumeral osteoarthritis, full thickness tears of the labrum or rotator cuff, tendinosis, calcific tendonitis)
* A history of significant trauma to the shoulder
* Poorly controlled diabetes mellitus, as defined by HbA1c > 7.5 mmol/L and glucose > 200 mg/dL. For diabetic participants HbA1c and glucose levels will be measured prior to intervention and documented for later analysis. For non-diabetic participants, previous labs will be utilized. All other medical diseases will be documented for later analysis.
* History of Cardiovascular Accident (CVA) such as stroke or Transient Ischemic Attack (TIA)
* Blood dyscrasias
* Use of any NSAIDs besides Tylenol. A letter will be sent to each participant's primary care physician(s) requesting that no additional pain medications be given for the duration of the study
* Prior shoulder surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Change in Pain as assessed by the Shoulder Pain and Disability Index (SPADI) | Baseline
  SPADI is a self-administered questionnaire that measures a combination of pain and functional disability. SPADI is scored from 0 to 100 with a high score representing more pain and disability.
Change in Pain as assessed by the Shoulder Pain and Disability Index (SPADI) | 4 weeks following injection
  SPADI is a self-administered questionnaire that measures a combination of pain and functional disability. SPADI is scored from 0 to 100 with a high score representing more pain and disability.
Change in Pain as assessed by the Shoulder Pain and Disability Index (SPADI) | 12 weeks following injection
  SPADI is a self-administered questionnaire that measures a combination of pain and functional disability. SPADI is scored from 0 to 100 with a high score representing more pain and disability.
Change in Pain as assessed by the Shoulder Pain and Disability Index (SPADI) | 6 months following injection
  SPADI is a self-administered questionnaire that measures a combination of pain and functional disability. SPADI is scored from 0 to 100 with a high score representing more pain and disability.

SECONDARY OUTCOMES:
Change in pain intensity as assessed by the Visual Analog Scale (VAS) | Baseline
  VAS is scored on a 100mm horizontal line that represents pain intensity, from 0mm to 100mm, with a higher score corresponding to increased pain intensity.
Change in pain intensity as assessed by the Visual Analog Scale (VAS) | 4 weeks following injection
  VAS is scored on a 100mm horizontal line that represents pain intensity, from 0mm to 100mm, with a higher score corresponding to increased pain intensity.
Change in pain intensity as assessed by the Visual Analog Scale (VAS) | 12 weeks following injection
  VAS is scored on a 100mm horizontal line that represents pain intensity, from 0mm to 100mm, with a higher score corresponding to increased pain intensity.
Change in pain intensity as assessed by the Visual Analog Scale (VAS) | 6 months following injection
  VAS is scored on a 100mm horizontal line that represents pain intensity, from 0mm to 100mm, with a higher score corresponding to increased pain intensity.
Change in range of motion as assessed by the Passive Range of Motion (PROM) assessment using a goniometer (left side) | Baseline
  A goniometer will be used to measure range of motion during the PROM assessment. The goniometer measures the angle between the beginning position and the ending position of available motion, and the result is reported in degrees.
Change in range of motion as assessed by the Passive Range of Motion (PROM) assessment using a goniometer (left side) | 4 weeks following injection
  A goniometer will be used to measure range of motion during the PROM assessment. The goniometer measures the angle between the beginning position and the ending position of available motion, and the result is reported in degrees.
Change in range of motion as assessed by the Passive Range of Motion (PROM) assessment using a goniometer (left side) | 12 weeks following injection
  A goniometer will be used to measure range of motion during the PROM assessment. The goniometer measures the angle between the beginning position and the ending position of available motion, and the result is reported in degrees.
Change in range of motion as assessed by the Passive Range of Motion (PROM) assessment using a goniometer (left side) | 6 months following injection
  A goniometer will be used to measure range of motion during the PROM assessment. The goniometer measures the angle between the beginning position and the ending position of available motion, and the result is reported in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Eric F Berkman, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No